CLINICAL TRIAL: NCT01996748
Title: A Multicenter, Randomized, Parallel, Double-blind, Clinical Trial Study to Assess the Efficacy and Safety of DF277 Compared to Placebo in Patients With Otic Eczema
Brief Title: Clinical Study to Assess the Efficacy and Safety of DF277 Compared to Placebo in the Treatment of Otic Eczema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF277OTIII/11ES01
Record Dates: First submitted 2013-10-14; First posted 2013-11-27 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Otic Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DF277 (Experimental): Two administrations daily for 7 days
  Interventions: Drug: DF277
- Placebo (Placebo Comparator): Two administrations daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DF277 — Two administrations daily for 7 days
  Arms: DF277
Drug: Placebo — Two administrations daily for 7 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of DF277 for the treatment of otic eczema.

ELIGIBILITY:
Inclusion Criteria:

* 12 years or older
* Clinical diagnosis of otic eczema suitable for local treatment

Exclusion Criteria:

* Other diseases.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorios SALVAT, S.A., Esplugues de Llobregat, Barcelone, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DF277 | Placebo
Started | 66 | 69
Completed | 58 | 63
Not Completed | 8 | 6
Not completed — Personal reason | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DF277 | Placebo | Total
Number analyzed (Participants) | 66 | 69 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 57 | 109
  >=65 years | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (12.7) | 52.2 (11.9) | 52.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 61 | 109
  Male | 18 | 8 | 26
Region of Enrollment [Number; unit: participants]
  Spain | 66 | 69 | 135

OUTCOME MEASURES:

1. Primary Outcome: Analysis of the Itching Change at the End of Treatment.
Description: The analysis of the itching change at the end of treatment (mean itching on days 4-8 compared to baseline). Itching was assessed on a 4 point ordinal scale; 0=absent, 1=mild, 2=moderate, 3=severe
Time Frame: Baseline and days 4-8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DF277 | Placebo
Number analyzed (Participants) | 66 | 69
units on a scale | -1.63 (0.82) | -1.25 (0.72)

2. Secondary Outcome: Change in Signs/ Symptoms
Description: - Change in itching at follow-up (mean itching on days 9-15 compared to baseline).
Time Frame: Baseline and days 9-15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DF277 | Placebo
Number analyzed (Participants) | 66 | 69
units on a scale | -1.80 (0.81) | -1.32 (0.77)

3. Secondary Outcome: Change in Mean Global Scores of Otoscopic Signs (Erythema, Edema and Scaling) at the End of Treatment (Day 8) Compared to Baseline (Day 1).
Description: Analysis of the change on global scores of otoscopic signs at the end of treatment (mean global scores of otoscopic signs on day 8 compared to baseline).
  Erythema, edema and scaling were assessed on a 4 point ordinal scale; 0=absent, 1=mild, 2=moderate, 3=severe.
Time Frame: Baseline and day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DF277 | Placebo
Number analyzed (Participants) | 66 | 69
units on a scale | -1.21 (0.68) | -0.78 (0.68)

4. Secondary Outcome: Change in Mean Global Scores of Otoscopic Signs (Erythema, Edema and Scaling) at the End of Follow-up (Day 15) Compared to Baseline (Day 1).
Description: Analysis of the change on global scores of otoscopic signs at the end of treatment (mean global scores of otoscopic signs on day 15 compared to baseline).
  Erythema, edema and scaling were assessed on a 4 point ordinal scale; 0=absent, 1=mild, 2=moderate, 3=severe.
Time Frame: Baseline and day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DF277 | Placebo
Number analyzed (Participants) | 66 | 69
units on a scale | -1.20 (0.68) | -0.77 (0.72)

ADVERSE EVENTS:
Time Frame: During all the study (15 days)
Arm/Group | DF277 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/69
Other Adverse Events (participants affected / at risk) | 4/66 | 10/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF277 (N=66) | Placebo (N=69)
Ear discomfort (Ear and labyrinth disorders) | 4 (5) | 5 (5)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not object to publication by Institution of the results of the Trial based on information collected or generated by Institution, whether or not the results are favorable to the Sponsor Drug. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Institution will provide Sponsor an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.